CLINICAL TRIAL: NCT04401644
Title: Laser Interferometry of Single Virus Particles Flowing Through Glass Microcapillaries to Detect Novel Coronavirus COVID-19
Brief Title: COVID-19: Laser Interferometry for Rapid Single Coronavirus Detection
Acronym: COLIDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Somerset NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other); University of Plymouth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBA20203
Record Dates: First submitted 2020-05-15; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Diagnoses Disease; Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: within group comparison of methods of detection of virus by two test methodologies. Post hoc validation of test performance against reference set.
Masking Description: The participants and the primary care provider will be masked to the outcome of the test. The test will not be used to determine clinical care and the result of the original diagnostic test will be masked from the outcomes assessor of the novel test under investigation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- primary arm (Experimental): There will only be one set of participants with each participants samples and results as the comparator groups. There will be within group comparison of methods of detection of virus by two test methodologies. Post hoc validation of test performance against reference set.
  Interventions: Diagnostic Test: Novel laser inferometry test for CORONA virus

INTERVENTIONS:
Diagnostic Test: Novel laser inferometry test for CORONA virus — detection of virus particles by light absorbtion patterns.

SUMMARY:
Using Laser light to detect COVID 19 virus particles in deep throat swab / nasal swab samples.

DETAILED DESCRIPTION:
The investigators will develop novel primers to detect single virus particles in patient samples. The method involves the absorption of light by single virus particles giving a specific pattern. The investigators will develop the device to create a microdroplet of carrier fluid that is run through the trial device. The investigators will develop novel binding receptors for preferential capture of Coronavirus.

The investigators will review the results of the novel test against the standard diagnostic test and identify virus particles in test negative subjects.

The investigators will isolate the viral rna in test negative subjects and perform sequencing to find novel mutations that are not detected by the current test.

ELIGIBILITY:
Inclusion Criteria:

* clinical suspicion of coronavirus or staff member having a coronavirus test

Exclusion Criteria:

* unable to give written informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
kappa value | 6 months
  level of agreement between novel test and standard test

SECONDARY OUTCOMES:
sensitivity and specificity | unknown this will require a centrally validated test set for known positives and negatives to be available estimated 1 year
  test of accuracy for the result versus a validated sample set

OTHER OUTCOMES:
clinical utility of test | 3 months
  timeliness of results

CONTACTS AND LOCATIONS:
Locations (1):
- Somerset NHS Foundation Trust, Taunton, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: No
During the trial, the investigators will store a list of participants and their unique trial number on a password protected file and computer in the Clinical Research Department. After the trial has completed, and when the data is stored or used, any information that could identify an individual participant will be removed or "pseudonymised". A pseudonym is a unique identifier which does not reveal the participant's 'real world' identity.
  Personal identifiable data will not be shared with any other outside organisation. The results of the tests will be shared with the collaborators using a unique trial number. Any remaining blood sample material will be frozen and stored as serum using the unique trial number in Musgrove Park Hospital's research laboratory.